CLINICAL TRIAL: NCT01066988
Title: Evaluation of an Investigational Lubricant Eye Drop on Lipid Layer Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-046
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: lipid layer thickness
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricants; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right Eye (Other): ORB Ocular Emulsion or SootheXP
  Interventions: Other: ORB Ocular Emulsion
- Left Eye (Other): ORB Ocular Emulsion or SootheXP
  Interventions: Other: SootheXP Emollient (Lubricant) Eye Drops

INTERVENTIONS:
Other: ORB Ocular Emulsion — lubricant eye drop
  Arms: Right Eye
Other: SootheXP Emollient (Lubricant) Eye Drops — lubricant eye drop
  Arms: Left Eye

SUMMARY:
The purpose of this study is to evaluate the effects of an investigational lubricant eye drop on tear film lipid layer thickness of dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (minimum age 18) meeting specific criteria for dry eye.

Exclusion Criteria:

* Use of topical ocular drops within 12 hours of the study visit; or use of topical ocular ointment within 36 hours of the study visit. In addition, cannot use any topical ocular drugs during study period.
* History or evidence of ocular or systemic medical conditions and/or medications that would confound the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Lipid layer thickness | Baseline through 120 minutes post instillation

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

REFERENCES:
- [Result] Benelli U. Systane lubricant eye drops in the management of ocular dryness. Clin Ophthalmol. 2011;5:783-90. doi: 10.2147/OPTH.S13773. Epub 2011 Jun 10. PMID 21750611